CLINICAL TRIAL: NCT00818246
Title: Non-ablative Light Source for the Treatment of Rhytides (Wrinkles)
Brief Title: Light Emitting Diode (LED) for the Treatment of Wrinkles
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: RoseLab Skin Optics Laboratory (Other)
Responsible Party: Dr Daniel Barolet, RoseLab Skin Optics Laboratory
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: LEDP-1
Record Dates: First submitted 2008-12-03; First posted 2009-01-07 (Estimated); Results first posted 2009-11-16 (Estimated); Last update posted 2009-11-16 (Estimated); Status verified 2009-10

CONDITIONS: Skin Aging; Photoaging of Skin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham light (Sham Comparator): one side of the face was treated three times weekly for four consecutive weeks (12 treatments) with a Sham light on the experimental periorbital area
  Interventions: Device: Sham light
- LED-treated (Experimental): one side of the face was treated three times weekly for four consecutive weeks (12 treatments) with 660 nm Light emitting diode (LED) on the experimental periorbital area
  Interventions: Device: LumiPhase-R™, OPUSMED Inc. Montreal, Canada

INTERVENTIONS:
Device: Sham light
  Arms: Sham light
Device: LumiPhase-R™, OPUSMED Inc. Montreal, Canada — 660 nm wavelength delivered in a sequential pulsing mode
  Arms: LED-treated

SUMMARY:
The purpose of this study was to determine whether light emitting diode (LED) therapy can improve skin appearance of human subjects with aged/photoaged skin. A reduction in rhytid depth as well as in skin surface roughness and in the degree of elastosis after LED treatments was expected.

ELIGIBILITY:
Inclusion Criteria:

* subjects with aged/photodamaged skin

Exclusion Criteria:

* Subjects were not allowed to participate in this study if they were taking cortisone (Prednisone), anticoagulant therapy, or any drug known to increase photosensitivity. In addition, during the 12 months preceding the study, subjects were required not to have used isotretinoin (Accutane), or applied topical steroids to the site to be treated. Moreover, previous laser or topical medication at the to-be-treated site was not permitted.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- RoseLab Skin Optics Laboratory, Montreal, Quebec, Canada

REFERENCES:
- [Result] Barolet D, Roberge CJ, Auger FA, Boucher A, Germain L. Regulation of skin collagen metabolism in vitro using a pulsed 660 nm LED light source: clinical correlation with a single-blinded study. J Invest Dermatol. 2009 Dec;129(12):2751-9. doi: 10.1038/jid.2009.186. Epub 2009 Jul 9. PMID 19587693

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham-treated; LED-treated (Split-face Study): one side of the face was treated with a Sham light and the other half with a light emitting diode (LED) at 660 nm three times weekly for four consecutive weeks (12 treatments)on the experimental periorbital area.
Period: Overall Study
Arm/Group | Sham-treated; LED-treated (Split-face Study)
Started | 40
Completed | 35 (split-face study)
Not Completed | 5
Not completed — Impossible to match pictures | 5

BASELINE CHARACTERISTICS:
Arm/Group | Sham-treated; LED-treated (Split-face Study)
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 3
Region of Enrollment [Number; unit: participants]
  Canada | 40

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Microtopographic Profilometry Ra Values (Skin Roughness).
Description: Phaseshift Rapid In vivo Measurement Of Skin (PRIMOS) readings. Analysis of the data in the image is used to generate Microtopographic profilometry Ra values (skin surface roughness).
Time Frame: Baseline and 4 weeks
Population: Per Protocol
Measure: Mean (95% Confidence Interval); unit: Percent change post-treatment
Arm/Group | Sham-treated; LED-treated (Split-face Study)
Number analyzed (Participants) | 35
Percent change post-treatment
  Sham-treated | 3.62 [-0.16 to 7.41]
  LED-treated | 18.57 [14.78 to 22.36]
Statistical Analysis 1: Comparison: Sham-treated; LED-treated (Split-face Study); Sample sizes and power calculations were generated according to the primary outcome measures of the study. In order to have a 98% chance of detecting as significant (at the two sided 5% level) a 10% difference between the treated and untreated/control sides in the Ra and Rz post-treatment improvement, with an assumed standard deviation of 10, 33 subjects were required. To account for an 80% per protocol completion rate, the planned number of patients to be enrolled was 40; Test type: Superiority or Other; p < 0.0001, ANCOVA; analysis of covariance (ANCOVA) was used to assess statistical differences between the LED-treated and untreated sides taking into account Age; Mean Difference (Final Values) = 14.94, Standard Error of Mean 2.68

2. Secondary Outcome: Change From Baseline in Units on the Fitzpatrick Classification System (FCS) Scale for Degree of Wrinkling.
Description: Clinical qualitative assessment was performed by three blinded medical observers through the evaluation of digital photographs. The photographs were analyzed for clinical improvement using the Fitzpatrick Classification System (FCS)subtype scale for degree of wrinkling (rhytids). Their assessment was rated on a five-point scale and scored as follows; 0=none; 1=mild; 2=moderate; 3=good; 4=excellent.
Time Frame: Baseline and 4 weeks
Population: Per Protocol
Measure: Mean (95% Confidence Interval); unit: Change in units on the FCS scale
Arm/Group | Sham-treated; LED-treated (Split-face Study)
Number analyzed (Participants) | 40
Change in units on the FCS scale
  Sham-treated | 0.48 [0.35 to 0.61]
  LED-treated | 1.08 [0.96 to 1.21]
Statistical Analysis 1: Comparison: Sham-treated; LED-treated (Split-face Study); Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.605, Standard Error of Mean 0.09

3. Primary Outcome: Percent Change From Baseline in Microtopographic Profilometry Rz Values (Rhytid Depth and Severity.
Description: Phaseshift Rapid In vivo Measurement Of Skin (PRIMOS) readings. Analysis of the data in the image is used to generate Microtopographic profilometry Rz values (peak to valley analysis) to quantify rhytid depth and severity.
Time Frame: Baseline and 4 weeks
Population: Per Protocol
Measure: Mean (95% Confidence Interval); unit: Percent change post-treatment
Arm/Group | Sham-treated; LED-treated (Split-face Study)
Number analyzed (Participants) | 35
Percent change post-treatment
  Sham-treated | 7.34 [3.37 to 11.31]
  LED-treated | 20.82 [16.85 to 24.79]
Statistical Analysis 1: Comparison: Sham-treated; LED-treated (Split-face Study); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 13.4, Standard Error of Mean 2.8

4. Secondary Outcome: Number of Adverse Events.
Description: Signs of erythema, edema, scaling/crusting, bronzing, textural changes, hyperpigmentation, and hypopigmentation were monitored.
Time Frame: Adverse reactions were monitored throughout the study and up to 4 weeks.
Population: Intention to treat (ITT)
Measure: Number; unit: Number of adverse events
Arm/Group | Sham-treated; LED-treated (Split-face Study)
Number analyzed (Participants) | 40
Number of adverse events
  Sham-treated | 0
  LED-treated | 0

ADVERSE EVENTS:
Arm/Group | Sham-treated; LED-treated (Split-face Study)
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes